CLINICAL TRIAL: NCT04367922
Title: A Positive Affect Regulation sKills Intervention to Decrease Stress During a Pandemic: A Single Arm, Non-Randomized Trial of a Public Platform
Brief Title: Positive Affect Regulation sKills at Northwestern University
Acronym: PARK-NU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00212262
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Anxiety; Depression; Social Isolation
MeSH Terms: conditions — Anxiety Disorders; Depression; Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive emotion skills invervention (Experimental): Participants will go through a 6-week positive emotion skills course where 1 new skill opens each week.
  Interventions: Behavioral: Positive Emotion Skills Course

INTERVENTIONS:
Behavioral: Positive Emotion Skills Course — The skills will be delivered over approximately 6 weeks, and individuals can participate from any device and location with internet access. A week will consist of 1-2 days of didactic material and 5-6 days of real-life skills practice and reporting. Participants cannot skip ahead, and can only progress to the next lesson if they have completed the current one, but they can return to old lessons or exercises if they wish to. Skills include: positive events, capitalizing, gratitude, mindfulness, positive reappraisal, personal strengths, achievable goals, self-compassion.

SUMMARY:
The Positive Affect Regulation sKills (PARK) Course is an online program containing a series of positive emotion skills for individuals experiencing stress and distress as a result of COVID-19 and the return to "normal." The study specifically targets positive emotion, and offers an array of skills in a self-guided online delivery platform, making the program accessible and convenient in confusing and stressful times.

Our main aims are:

Aim 1: To explore the effects of PARK on anxiety, depression, feelings of social isolation, positive affect, and a sense of meaning and purpose.

Aim 2: To test whether age or gender moderate the effects of the program.

DETAILED DESCRIPTION:
The goal of the proposed program, PARK, is to reduce feelings of anxiety, depression, and social isolation, as well as increase well-being and a sense of meaning and purpose through the practice of positive emotion skills via a self-guided online platform. We will compare baseline scores on PROMIS measures of Anxiety, Depression, Social Isolation, Meaning and Purpose, and Positive Emotion to scores after completing the online course (approximately 8 weeks later), and again at 6 months post-baseline.

Research will be based in Northwestern's Feinberg School of Medicine through the Department of Medical Social Sciences (MSS), with all study procedures conducted online. Eligibility screening, consent, and assessments will be conducted on REDCap. For the positive skills course (including weekly lessons and daily skills practice) and daily emotion check-ins, consenting participants will receive access to the online PARK platform, hosted by BrightOutcome.

The skills will be delivered over approximately 6 weeks, and individuals can participate from any device and location with internet access.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Speaks and reads English
* Able to access the online platform through their phone, a public device (i.e., at the library) or at home.
* Lives in US

Exclusion Criteria:

* Inability to communicate in English
* Lives outside the US
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | Baseline, 6 weeks, 6 months
  Assessed using PROMIS Anxiety (CAT)
Change in depression | Baseline, 6 weeks, 6 months
  Assessed using PROMIS Depression (CAT)
Change in feelings of social isolation | Baseline, 6 weeks, 6 months
  Assessed using PROMIS Social Isolation (CAT)
Change in positive affect | Baseline, 6 weeks, 6 months
  Assessed using PROMIS Positive Affect (CAT)
Change in sense of meaning and purpose | Baseline, 6 weeks, 6 months
  Assessed using PROMIS Meaning and Purpose (CAT)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Moskowitz, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moskowitz JT, Addington EL, Cheung EO. Positive psychology and health: Well-being interventions in the context of illness. Gen Hosp Psychiatry. 2019 Nov-Dec;61:136-138. doi: 10.1016/j.genhosppsych.2019.11.001. Epub 2019 Nov 8. No abstract available. PMID 31757566
- [Background] Addington EL, Cheung EO, Bassett SM, Kwok I, Schuette SA, Shiu E, Yang D, Cohn MA, Leykin Y, Saslow LR, Moskowitz JT. The MARIGOLD study: Feasibility and enhancement of an online intervention to improve emotion regulation in people with elevated depressive symptoms. J Affect Disord. 2019 Oct 1;257:352-364. doi: 10.1016/j.jad.2019.07.049. Epub 2019 Jul 5. PMID 31302525
- [Background] Moskowitz JT, Cheung EO, Snowberg KE, Verstaen A, Merrilees J, Salsman JM, Dowling GA. Randomized controlled trial of a facilitated online positive emotion regulation intervention for dementia caregivers. Health Psychol. 2019 May;38(5):391-402. doi: 10.1037/hea0000680. PMID 31045422
- [Background] Bassett SM, Cohn M, Cotten P, Kwok I, Moskowitz JT. Feasibility and Acceptability of an Online Positive Affect Intervention for Those Living with Comorbid HIV Depression. AIDS Behav. 2019 Mar;23(3):753-764. doi: 10.1007/s10461-019-02412-z. PMID 30701389
- [Background] Pressman SD, Jenkins BN, Moskowitz JT. Positive Affect and Health: What Do We Know and Where Next Should We Go? Annu Rev Psychol. 2019 Jan 4;70:627-650. doi: 10.1146/annurev-psych-010418-102955. Epub 2018 Sep 27. PMID 30260746
- [Background] Cheung EO, Addington EL, Bassett SM, Schuette SA, Shiu EW, Cohn MA, Leykin Y, Saslow LR, Moskowitz JT. A Self-Paced, Web-Based, Positive Emotion Skills Intervention for Reducing Symptoms of Depression: Protocol for Development and Pilot Testing of MARIGOLD. JMIR Res Protoc. 2018 Jun 5;7(6):e10494. doi: 10.2196/10494. PMID 29871853
- [Background] Cohn MA, Pietrucha ME, Saslow LR, Hult JR, Moskowitz JT. An online positive affect skills intervention reduces depression in adults with type 2 diabetes. J Posit Psychol. 2014 Jan 1;9(6):523-534. doi: 10.1080/17439760.2014.920410. PMID 25214877
- [Background] Dowling GA, Merrilees J, Mastick J, Chang VY, Hubbard E, Moskowitz JT. Life enhancing activities for family caregivers of people with frontotemporal dementia. Alzheimer Dis Assoc Disord. 2014 Apr-Jun;28(2):175-81. doi: 10.1097/WAD.0b013e3182a6b905. PMID 24113564
- [Background] Folkman S, Moskowitz JT. Coping: pitfalls and promise. Annu Rev Psychol. 2004;55:745-74. doi: 10.1146/annurev.psych.55.090902.141456. PMID 14744233
- [Derived] Addington EL, Cummings P, Jackson K, Yang D, Moskowitz JT. Exploring Retention, Usage, and Efficacy of Web-Based Delivery of Positive Emotion Regulation Skills During the COVID-19 Pandemic. Affect Sci. 2022 Oct 4;4(1):118-130. doi: 10.1007/s42761-022-00135-4. eCollection 2023 Mar. PMID 36211530